CLINICAL TRIAL: NCT03958682
Title: Design and Application of Airborne Visual Real-time Evaluation System for Air Medical Rescue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: I2018001352
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Medical Emergencies
Keywords: air medical rescue; satellite information transmission; Augmented Reality

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): During the rescue, the doctor is asked to wear the special helmet , through the device's camera system and headset, we can obtain graphics and sound of the helicopter cabin .At the same time, it also receives the historical data of patients and real-time diagnosis as well as rescue guidance from the ground medical institutions.Patients can receive timely diagnosis and appropriate treatment
  Interventions: Device: AR smart wearing equipment combined with 4G + satellite information transmission system

INTERVENTIONS:
Device: AR smart wearing equipment combined with 4G + satellite information transmission system — We are going to add a pair of wearable smart glasses with AR function to the original flight helmet .During the rescue, the doctor is asked to wear the special helmet , through the device's camera system and headset, we can obtain graphics and sound of the helicopter cabin .At the same time, it also receives the historical data of patients and real-time diagnosis as well as rescue guidance from the ground medical institutions.
  It can not only transmit the patient's information in the cabin to the ground medical institutions in real time, but also transmit the rescue plan of the ground medical experts to the rescue helicopter in real time to ensure the safety of patients in transit ,which will save the time for medical staff to hand over after landing and reduce errors.

SUMMARY:
This study intends to use AR (Augmented Reality) smart wearing equipment combined with 4G + satellite information transmission system to achieve two-way real-time information transmission in air-to-ground medical rescue.

DETAILED DESCRIPTION:
Investigators are going to add a pair of wearable smart glasses with AR function to the original flight helmet .During the rescue, the doctors are asked to wear the special helmet, through the device's camera system and headset, investigators can obtain graphics and sound of the helicopter cabin .At the same time, it also receives the historical data of patients and real-time diagnosis as well as rescue guidance from the ground medical institutions.

In short ,it can not only transmit the patient's information in the cabin to the ground medical institutions in real time, but also transmit the rescue plan of the ground medical experts to the rescue helicopter in real time to ensure the safety of patients in transit ,which will save the time for medical staff to hand over after landing and reduce errors.

At present, most of the airborne information exchange systems in air medical rescue in China focus on the internal use of the army, which are incompatible with the medical information systems of most hospitals on the ground. Moreover, these systems can only achieve limited information transmission, and can not delivery rescue scene images in real time. Civil air medical rescue conditions are relatively backward, most of them rely on 2G/3G/4G mobile communication technology, which can lead to failure in case of bad weather or sudden major disasters, and bring great security risks to patients in air medical rescue.

If the airborne visual real-time evaluation system can be successfully completed, it will be popularized and applied in Chinese airborne first aid alliance, and eventually a standardized airborne medical rescue information management system will be formed. Furthermore, a three-dimensional rescue system for civil airborne medical rescue will be built to reduce the potential safety hazards of patients in airborne medical rescue, and to enhance the rapid response ability and organization of medical institutions.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients who require air transportation support;
* Patients informed consent and sign the informed consent form

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of data correctly transmitted | each rescue, for 1 year
  Record the data sent from the ground hospital or helicopter cabin and data received in the helicopter cabin or ground hospital. Calculate the percentage of correctly transmitted data.
Time-consuming | each rescue, for 1 year
  The time required for data transmission

SECONDARY OUTCOMES:
Satisfaction index | each rescue, for 1 year
  Design a questionnaire to evaluate the satisfaction of using the device by doctors and nurses. The questionnaire consists five items rating from 1 to 5. 1 represents extremely not satisfied, 5 represents very satisfied. The highest score is 25.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China